CLINICAL TRIAL: NCT07174934
Title: Evaluation of The Effect of Injectable Platelet-Rich Fibrin Application on Wound Healing Following Gingivectomy or Gingivoplasty: Randomized Controlled Clinical Study
Brief Title: Effect of I-PRF After Gingivectomy
Acronym: I-PRF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Eman Ahmed Elgharib Ahmed, Dentist at Egyptian Ministry of Health, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-ME-25-07
Record Dates: First submitted 2025-09-12; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: Chronic Inflammatory Gingival Enlargement

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Outcomes Assessor and Care Provider will be masked about type of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- application of injectable platelet-rich fibrin after gingivectomy or gingivoplasty . (Active Comparator): 10 systemically healthy patients with chronic inflammatory gingival enlargement will be randomly treated with gingivectomy or gingivoplasty and application of injectable platelet rich fibrin on wound area.
  Interventions: Biological: application of injectable platelet-rich fibrin on the wound area .
- gingivectomy or gingivoplasty alone (No Intervention): 10 systemically healthy patients with chronic inflammatory gingival enlargement will be randomly treated with gingivectomy or gingivoplasty alone (control).

INTERVENTIONS:
Biological: application of injectable platelet-rich fibrin on the wound area . — Injectable platelet-rich fibrin will be prepared using low speed centrifugation technique, after centrifugation, the I-PRF in the upper part of the tube will be collected via an injector and will be transferred to a metal godet. It will be left for 15-20 min for polymerization of the I-PRF ,Then the polymerized I-PRF will be applied to the secondary wound of test area.
  Arms: application of injectable platelet-rich fibrin after gingivectomy or gingivoplasty .

SUMMARY:
The goal of this clinical trial is to evaluate the effect of injectable platelet-rich fibrin application on wound healing following gingivectomy or gingivoplasty.

The main question it aims to answer are:

Does the injectable platelet-rich fibrin enhance the wound healing after gingivectomy or gingivoplasty ?

Participants(who have chronic inflammatory gingival overgrowth) will be divided into two groups :

Group I: systemically healthy patients with chronic inflammatory gingival enlargement will be randomly treated with gingivectomy or gingivoplasty alone (control).

Group II: systemically healthy patients with chronic inflammatory gingival enlargement will be randomly treated with gingivectomy or gingivoplasty and application of injectable platelet rich fibrin on wound area.

The patients will be recalled for follow-up appointments on days 7, 14, and 21.

DETAILED DESCRIPTION:
All participants will receive a full-mouth clinical examination, Initial periodontal therapy and oral hygiene instructions. the patients will be called again 2 weeks later after phase I therapy.

The following periodontal parameters will be recorded: Plaque Index (PI) , Bleeding on probing (BOP) before and after surgery operation at (baseline, 21day).

Prior to the procedure, patients will be rinsed with mouthwash containing 0.12% chlorhexidine. Surgical operations will be carried out with local infiltration anesthesia with vasoconstrictor the gingivectomy or gingivoplasty operation will be done with the conventional method (the procedure of gingivectomy with a #15 scalpel), then Test group: I-PRF is placed on the wound area after a gingivectomy or gingivoplasty with the conventional method and closed with a periodontal dressing.

Control group: closure of the wound area with only a periodontal dressing after a gingivectomy or gingivoplasty with the conventional method.

Post-operative instructions will be given and patients will be asked to avoid brushing at the surgical sites for at least 7 days, 0.2% chlorhexidine gluconate mouthwash twice daily for 14 days will be prescribed.

Clinical follow-up of patients:

The patients will be recalled for follow-up appointments on days 7, 14, and 21. The parameters evaluated in the control sessions were as follows:

1. LTH wound healing index : there are many parameters to assess wound healing, but the Landry, Turnbull, and Hawley Index is easy and convenient to score . It has a scoring range from 1 to 5, the lowest being 1 and the highest being 5. The parameters measured in this index are the healing index, tissue color, bleeding on palpation, granulation tissue, and suppuration .
2. MMS scale : the modified Manchester scar scale (MSS) was used to assess the color, contour, and distortion of the wound .

   The color of the wound was classified as a perfect match (score 0), mild mismatch (score 1), or obvious mismatch (score 2) compared with the neighboring mucosa. The contour of the wound was evaluated as similar (score0), slightly raised, or indented (score 1) and hypertrophic (score2) when compared with surrounding tissues. Wound distortion was evaluated as no distortion (score 0), mild distortion (score 1), and obvious distortion (score 2). The sum of the scores in the three categories shows the repair score of the wound, with a total score ranging from 0 to 6, with lower scores indicating better repair.
3. Visual Analog Scale : Assessment patient satisfaction very important so, post operative pain will be evaluated by visual analog scale (VAS) . In this method, the patients will be asked to rate their pain at an examination in form of a score between 0 (no pain) and 100 (the most pain which patient has ever experienced) .

Gingival fluid sampling :

Gingival crevicular fluid (GCF) collection will be done before the operation (at base line), and after the operation (21th day). samples will be collected using sterile paper strips, Paper strips contaminated with blood or saliva will be discarded.

The samples will be assayed for PRL by using an enzyme linked immunosorbent assay (ELISA) kits.

full-mouth clinical examination, Initial periodontal therapy, clinical measurements, surgery operation, gingival crevicular fluid sampling and follow-up evaluations will be performed by the same periodontist.

ELIGIBILITY:
Inclusion Criteria:

* 1- Systemically healthy patients. 2- patients ages18-35years. 3- patients with chronic inflammatory gingival overgrowth. 4- patients with fibrotic gingival overgrowth. 5- Patients with enough attached gingiva. 6- Patients signing informed written consent.

Exclusion Criteria:

- 1) Pregnancy or lactation. 2) Any known systemic disease. 3) Any type of previous periodontal treatment (surgical or non-surgical) in the preceding 6 months.

4) smokers and alcohol users 5) clinical attachment or bone loss. 6) Patients run on immunosuppressive agents, systemic corticosteroids, chemotherapy, and/or radiotherapy drugs taken or prescribed 2 months before the study attempt, which may affect the study results, wound healing, and coagulation mechanism.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in gingival crevicular fluid level of Vascular Endothelial Growth Factor (VEGF) at baseline and 21 days after gingivectomy or gingivoplasty. | at baseline, 21days after gingivectomy.

SECONDARY OUTCOMES:
Patient satisfaction using Visual Analog Scale (VAS). | At 7th ,14th,21th days after gingivectomy.
  Scale Range: 0 (not satisfied at all) to 10 (completely satisfied).
Clinical wound healing using Landry, Turnbull, and Howley (LTH) Wound Healing Index. | 7th, 14th, 21st days after gingivectomy.
  Scale Range: 1 (very poor healing) to 5 (excellent healing).
Clinical wound healing using Modified Manchester Scar (MMS) Scale. | 7th, 14th, 21st days after gingivectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Out-Patient Clinic of Oral Medicine, Periodontology, Oral Diagnosis and Radiology department, Faculty of Dental Medicine for Girls, Al-Azhar University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No